CLINICAL TRIAL: NCT05461001
Title: Effects of Sport-specific Endurance Running on Cardiorespiratory Fitness in Football Players
Brief Title: Sport-specific Endurance Training on Cardiorespiratory Fitness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0406 Maria
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cardiorespiratory Fitness
Keywords: sport specific endurance
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Up Exercises daily for Cardiorespiratory Fitness (Experimental): Effect of warm up activities daily on cardiorespiratory fitness of Male Football Players
  Interventions: Other: Warm Up Exercises
- Endurance based Exercises for Cardiorespiratory Fitness (Experimental): Effect of sports-specific endurance based exercises on cardiorespiratory fitness of Male Football Players
  Interventions: Other: Endurance Based Exercises

INTERVENTIONS:
Other: Warm Up Exercises — The daily warm up exercises for male football players include full body stretch, high knees, lunges, squat and burpees.
  Arms: Warm Up Exercises daily for Cardiorespiratory Fitness
Other: Endurance Based Exercises — Sport-specific endurance-running (duration [in minutes], total distance [in meters], mean speed [in meters per minute], high-speed running >15 km·h-1, and relative high-speed running [>75% and >85% of maximal velocity]) will be given to the experimental group. Athletes will run in excess of 15 km of total distance (TD) and 4 km of high-speed (>15 km·h-1) distance per session 3 to 4 running-based endurance sessions per week for 6 weeks.
  Arms: Endurance based Exercises for Cardiorespiratory Fitness

SUMMARY:
The football players require a number attributes for excellent performance. These attributes include cardiovascular fitness, muscle strength, muscular Endurance, flexibility, agility, Coordination, skill and tactical knowledge. In young male football players, the most important attributes are high levels of skill in passing, shooting, dribbling, and heading. A long-term commitment to endurance training is necessary to reach and maintain a player full physical potential. There are two primary objectives of the endurance program are to prevent injury and enhance the abilities to play the game.

DETAILED DESCRIPTION:
The football players require a number attributes for excellent performance. These attributes include cardiovascular fitness, muscle strength, muscular Endurance, flexibility, agility, Coordination, skill and tactical knowledge. In young male football players, the most important attributes are high levels of skill in passing, shooting, dribbling, and heading. A long-term commitment to endurance training is necessary to reach and maintain a player full physical potential.

In sport-specific endurance running on cardiorespiratory fitness endurance, 26 male football players with age group of 16-25 are selected. The participants have never undergone surgery or accident and do not possess any lethal disease. The participants will be allocated into control group with 13 participants and experimental group with 13 participants respectively. The sample will be taken in study setting of Pakistan Sports Board. Control group will follow their daily warm up activities. Interventional group will follow the endurance-based running protocol. Sport-specific endurance-running (duration [in minutes], total distance [in meters], mean speed [in meters per minute], high-speed running >15 km·h-1, and relative high-speed running [>75% and >85% of maximal velocity]) will be given to the experimental group. Athletes will run in excess of 15 km of total distance (TD) and 4 km of high-speed (>15 km·h-1) distance per session 3 to 4 running-based endurance sessions per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male Football players
* Age Group: 16-25 years
* Already working on endurance based exercises

Exclusion Criteria:

* Female Football players
* Players undergone surgery or accident
* Any malignant disease or chronic disease

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 24 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Cooper Test | 6 week
  Participants started running on athletics track. The subjects did their best to run many laps around running track for 12 minutes. When 12 minutes over the subjects stopped running and they stood on their spot. Then, the amount of distance covered by subjects within twelve minutes and the exercise heart rate (EHR) of each subject were measured in meter and beat per minute. In addition, after getting plenty of resting time, resting heart rate (RHR) of the subjects was measured in best minute
Shuttle Run | 6 week
  For assessment of speed and agility, the shuttle run test (10 × 5m) was applied. Shuttle runs are a popular training technique for sports which involve short bursts of speed. They help develop your acceleration, speed and your anaerobic fitness. In shuttle run, the participant run to the 10m mark first, touching the floor and running back to the start line. Then run to the 20m line and back. Finally run to the 30m line and back. Start the routine again and repeat four times
Indirect VO2 Calculation | 6 week
  The VO2 maximum of male football players is calculated using formula

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Borad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No